CLINICAL TRIAL: NCT02458586
Title: Ernährungs-Interventions-Fettleber-Studie (Interventional Study on Nutritional Effects on NAFLD)
Acronym: UFOP-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: ufop: Union zur Förderung von Oel- und Proteinpflanzen e.V. (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Head of Department of Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFOP-2
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: NAFLD; Obesity; Prediabetes; Dyslipoproteinemia
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Prediabetic State; Dyslipidemias | interventions — Diet Therapy; Counseling

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MUFA (Placebo Comparator): daily intake of 50 g of olive oil over a period of 8 weeks
  Interventions: Dietary Supplement: Dietary intervention / counseling
- PUFA (Active Comparator): daily intake of 50 g of canola oil (rapeseed oil) over a period of 8 weeks
  Interventions: Dietary Supplement: Dietary intervention / counseling

INTERVENTIONS:
Dietary Supplement: Dietary intervention / counseling — dietary counseling and daily intake of 50 g of dietary oil over a period of 8 weeks

SUMMARY:
Epidemiological data and studies in animal models suggest, that polyunsatured fatty acids (PUFA) rather than mono-unsatured fatty acids (MUFA) are associated with lower hepatic lipid content (HCL) and may facilitate a decrease of HCL in case of non-alcoholic fatty liver disease (NAFLD).

The investigators therefore conduct an interventional trial in subjects with normal glucose metabolism, but increased HCL, fulfilling criteria for NAFLD.

The study will compare two dietary interventions in parallel design, one containing mainly PUFA (canola oil), one containing only MUFA (olive oil). The intervention of 8 weeks is accomodated by dietary counseling. Metabolic outcome variables will be assessed with MR spectroscopy (liver fat) and euglycemic hepatic clamp (glucose metabolism/insulin sensitivity).

DETAILED DESCRIPTION:
Epidemiological data and studies in animal models suggest, that polyunsatured fatty acids (PUFA) rather than mono-unsatured fatty acids (MUFA) are associated with lower hepatic lipid content (HCL) and may facilitate a decrease of HCL in case of non-alcoholic fatty liver disease (NAFLD). A typical source for PUFAs are fish and certain plant oils, a source of almost pure MUFAs is olive oil.

The investigators therefore conduct an interventional trial in subjects with normal glucose metabolism, but increased HCL, fulfilling criteria for NAFLD. The investigation focusses on male participants to avoid sex-related differences in the results.

The study will compare two isocaloric dietary interventions in parallel design, one containing mainly PUFA (canola oil), one containing only MUFA (olive oil). The intervention of 8 weeks is accomodated by dietary counseling (4 sessions). Metabolic outcome variables will be assessed with MR spectroscopy (liver fat), anthropometry (to check for stable weight and body composition) and euglycemic hepatic clamp (glucose metabolism/insulin sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* increased hepatic fat content (NAFLD)
* BMI between 30 and 35 kg/m²

Exclusion Criteria:

* diabetes
* severe cardiac, pulmonary or gastrointestinal disorders
* hepatic disorders other than NAFLD
* alcoholism
* medication with metabolic side or main effects (e.g. statins)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
change in liver fat content | 4 and 8 weeks
  change in liver fat content (MR spectroscopy and ultrasound)
change in hepatic insulin sensitivity | 8 weeks only
  change in hepatic insulin sensitivity (euglycemic hepatic clamp)

CONTACTS AND LOCATIONS:
Locations (1):
- German Institut for Human Nutrition; Department for Clinical Nutrition, Nuthetal, Brandenburg, Germany